CLINICAL TRIAL: NCT02654600
Title: Variations of the Lung Compliance During Extracorporeal Circulation and Post Operative Pulmonary Complications
Acronym: COMPLI
Status: Completed | Type: Observational
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: P14-37816002/2014-A00702-45
Record Dates: First submitted 2015-09-02; First posted 2016-01-13 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Thoracic Surgery; Cardiopulmonary Bypass
Keywords: cardiac surgery; thoracopulmonary compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
the decrease in thoracopulmonary compliance after cardiac surgery is well known . The investigators hypothesize that the major factor determining pulmonary outcome after cardiac surgery is the alteration of pulmonary compliance during cardiopulmonary bypass(CBP) and that this alteration is due to CBP itself through pulmonary blood emptying.

DETAILED DESCRIPTION:
compliance is the compliance calculate when thorax is closed, the pulmonary compliance is the compliance calculated when thorax is opened After operation chest X-ray are daily done and blood samples as needed. Were recorded death, time of extubation,duration of non invasive ventilation,of Intensive Care Unit stay and of total hospital stay, troponin peak, lactates, blood gases, ionogram and count.Variations of compliance is analyzed through one factor paired Anova or Wilcoxon paired test. Decrease of compliance and respiratory complications are analyzed through binomial logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for standard aortic
* mitral or coronary surgery

Exclusion Criteria:

* emergency operation
* no complete preoperative echocardiography
* surgery needing multiple table position changes
* unstable cardiac or respiratory condition
* difficult patient needing multiple care and/or special attention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every ASA 2 or 3 patient eligible for non-complex and non-urgent cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
pulmonary compliance during cardiac surgery | intraoperative
  compliance is calculated by dividing tidal volume (ml) by the difference between plateau-inspiratory pressure (mmHg) and end-expiratory pressure (mmHg) before ,during and after CBP

SECONDARY OUTCOMES:
pulmonary complications including death after cardiac surgery | 1 month
  intersticial and/or alveolar pulmonary oedema leading to death or extra hospital stay
thoracopulmonary compliance during cardiac surgery | intraoperative
  compliance is calculated by dividing tidal volume (ml) by the difference between peak-inspiratory pressure (mmHg) and end-expiratory pressure (mmHg) before ,during and after CBP

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France

REFERENCES:
- [Background] Ellison LT, Duke JF 3rd, Ellison RG. Pulmonary compliance following open-heart surgery and its relationship to ventilation and gas exchange. Circulation. 1967 Apr;35(4 Suppl):I217-25. doi: 10.1161/01.cir.35.4s1.i-217. No abstract available. PMID 6024032
- [Background] Suter PM, Fairley HB, Isenberg MD. Effect of tidal volume and positive end-expiratory pressure on compliance during mechanical ventilation. Chest. 1978 Feb;73(2):158-62. doi: 10.1378/chest.73.2.158. PMID 340159